CLINICAL TRIAL: NCT07125690
Title: Effect of Local Heat Application and Oral Sucrose Use Before Heel Pick Collection on Pain, Stress, and Procedure Duration in Newborns
Brief Title: Effect of Two Non-pharmacological Method on Pain, Stress Procedure Duration in Newborn
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: TC Erciyes University (Other)
Responsible Party: Principal Investigator, FATMA GUL TAMER, PhD student, TC Erciyes University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: ErciyesU.FGTamer.01
Record Dates: First submitted 2025-08-09; First posted 2025-08-15 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2023-12

CONDITIONS: Neonatal Pain; Non-Pharmacological Pain Management
Keywords: neonatal; procedural pain; heel lancing; local heat applications; oral sucrose
MeSH Terms: conditions — Pain, Procedural | interventions — Sucrose

STUDY DESIGN:
Intervention Model Description: The process will be explained using the consent forms distributed to births that meet the inclusion criteria, and written consent will be obtained from the families. A Newborn and Family Identifying Information Form was first completed for the babies to be included in the study.For all groups to be included in the study, before the heel blood was taken, the Newborn Infant Pain Scale (NIPS), ALPS-Neo and physiological parameters were recorded on video with the babies' entire bodies visible, starting 6 minutes before the procedure, continuing during the procedure and ending 2 minutes after the procedure.The heel prick blood collection procedure was performed by the same healthcare professional each time, with the babies in the same position, and the data collection was performed by the researcher.
Who Masked: Participant, Outcomes Assessor
Masking Description: During the application, the family of the participating newborns does not know which group they will be included in.
  Experts who used pain scales to evaluate the videos used during the application. And they did not know which group the newborn were in.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Local Heat Application to the Heel (Active Comparator): The newborns included in this group received local dry heat application 5 minutes before the heel prick procedure, with the newborn in the supine position. Local dry heat was applied using a thermometer heated with water between 40 and 45˚C. The temperature of the water inside the thermometer was measured before application. The thermometer was applied to the sole of the newborn's right foot. Contact with bare skin was prevented, and the thermometer was used in a protective cover.
  Interventions: Other: local heat application
- Oral Sucrose Administration (Active Comparator): In accordance with the Neonatal Pain and Treatment Guidelines, a total of 1 ml of sucrose at a 24% concentration recommended for full-term infants was prepared in a syringe. It was administered to the anterior tongue 2 minutes before the heel prick.
  Interventions: Other: oral sucrose
- Local Heat and Oral Sucrose Application to the Heel (Active Comparator): Newborns included in the combined intervention group received local dry heat with a thermometer heated with water at 40-45˚C 5 minutes before blood collection, with the infant in the supine position. At the third minute of the local heating, 1 ml of 24% sucrose was applied to the anterior tongue over 1 minute. A stopwatch was used to monitor the procedure times.
  Interventions: Other: mixed group

INTERVENTIONS:
Other: local heat application — The newborns included in this group received local dry heat application 5 minutes before the heel prick procedure, with the newborn in the supine position. Local dry heat was applied using a thermometer heated with water between 40 and 45˚C. The temperature of the water inside the thermometer was measured before application. The thermometer was applied to the sole of the newborn's right foot. Contact with bare skin was prevented, and the thermometer was used in a protective cover.
  Arms: Local Heat Application to the Heel
Other: oral sucrose — In accordance with the Neonatal Pain and Treatment Guidelines, a total of 1 ml of sucrose at a 24% concentration recommended for full-term infants was prepared in a syringe. It was administered to the anterior tongue 2 minutes before the heel prick
  Arms: Oral Sucrose Administration
Other: mixed group — Newborns included in the combined intervention group received local dry heat with a thermometer heated with water at 40-45˚C 5 minutes before blood collection, with the infant in the supine position. At the third minute of the local heating, 1 ml of 24% sucrose was applied to the anterior tongue over 1 minute. A stopwatch was used to monitor the procedure times.
  Arms: Local Heat and Oral Sucrose Application to the Heel

SUMMARY:
This study is planned as a prospective, single-blind, randomized controlled experimental study matched according to gestational age, gender, and birth weight, to determine the effects of local heat application and oral sucrose use during heel prick blood collection on pain, stress, procedure duration, and physiological parameters of newborns.

DETAILED DESCRIPTION:
Non-pharmacological methods are important alternatives for managing pain caused by minimally invasive procedures performed on newborns. Applying local heat to the heel, one of the non-pharmacological methods that can be used to reduce pain during heel prick in newborns, suppresses pain escalation by activating the gate-control mechanism, reduces pain, stimulates sensory receptors, and induces vasodilation. It also reduces ischemic pain, promotes the removal of metabolic waste, increases endorphin release, inhibits muscle contraction, reduces the effects of pressure, and provides pain relief for newborns.

Another non-pharmacological method used for pain management in newborns is oral sucrose administration. Used as an analgesic in minor invasive procedures, sucrose activates the endogenous opioid system by stimulating the sense of taste. Oral sucrose administration is an easily administered, proven, readily available, inexpensive, and rapidly effective method.

Authorities have an important role to play in minimizing the negative effects of various invasive procedures and cutting procedures, and protecting the baby from the short- and long-term effects of pain. Natural, economical, and easily curative methods for reducing pain during heel punctures include sucrose administration and topical heat application to the heel, among the herbal solutions offered by Mothers and Organics.Various non-pharmacological methods have been investigated in the literature for their effects on pain during heel prick blood sampling, and the positive effects of sucrose injection and heat application to the heel have also been reported. However, studies have generally focused on the use of sucrose injection and local heat application to the heel alone for pain reduction. There is no study evaluating their combined use in the same sample and comparing their effects.Therefore, this study aims to determine the effects of local heat application to the heel and oral sucrose administration during heel prick blood collection on the pain, stress, physiological parameters, and procedure duration of newborns.

ELIGIBILITY:
Inclusion Criteria:

* 38-42 weeks gestational age,
* birth weight ≥ 2500 g,
* stable vital signs,
* no congenital anomalies,
* no congenital illnesses at birth such as neonatal asphyxia, hemolytic status, metabolic disease, skin disease, patent ductus arteriosus (PDA), respiratory distress syndrome (RDS), and sepsis,
* no intracranial hemorrhage,
* not taking any medications other than antibiotics and vitamin supplements,
* not fed or changed within 30 minutes before the heel prick,
* not taking opioids or sedatives within 4 hours before the heel prick,
* not undergoing any painful procedures at least one hour before the heel prick,
* newborns whose mothers gave verbal and written informed consent

Exclusion Criteria:

* Newborns who exhibited signs of infection (gastroenteritis, sepsis, etc.) during the study,
* Blood collection was not possible on the first attempt,
* Newborns whose mothers wished to withdraw from the study

Ages: 3 Days to 31 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 100 (Actual)
Dates: Start 2023-12-11 (Actual); Primary Completion 2023-12-11 (Actual); Study Completion 2024-06-03 (Actual)

PRIMARY OUTCOMES:
ALPS-Neo Pain and Stress Assessment Scale | 6 month
  The ALP-Neo performance is a three-point Likert-type scale consisting of five items: the subject's facial expression, breathing pattern, extremity tone, hand and foot activity, and activity level. Measurements are made through observation. The resulting score reflects increased stress and pain (3-5 points = mild pain and stress; >5 points = severe pain and stress).
Newborn Infant Pain Scale (NIPS) | 6 month
  The scale consists of five behavioral parameters, including facial expression, crying, breathing pattern, arm and leg movements, and alertness, and one physiological parameter that tracks breathing pattern. Each behavior except crying is scored from 0 to 1, and the crying parameter is scored from 0, 1, and 2. The NIPS scores range from 0 to 7, with 0-2 indicating no pain, 3-4 indicating moderate pain, and >4 indicating severe pain. Cronbach's alpha coefficients for the scale were calculated as 0.95, 0.87, and 0.88 before, during, and after the intervention, respectively.

CONTACTS AND LOCATIONS:
Overall Officials: fatma gul tamer, Principal Investigator — TC Erciyes University
Locations (1):
- Erciyes University, Kayseri, Kayseri, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No